CLINICAL TRIAL: NCT04219956
Title: A Prospective Randomized Multicenter Study to Evaluate the Efficacy of a Polyamine-deficient Diet for the Treatment of Postoperative Pain After Abdominal Surgery.
Brief Title: Study to Evaluate the Efficacy of a Polyamine-deficient Diet for Treating Postoperative Pain After Abdominal Surgery
Acronym: POLYAMAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: Centre de Recherche en Nutrition Humaine Ouest (CRNH) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC19_0023
Record Dates: First submitted 2020-01-03; First posted 2020-01-07 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Digestive System Surgical Procedures
Keywords: Abdominal surgery; Polyamine; Postoperative pain; Morphine; Hypersensitivity
MeSH Terms: conditions — Pain, Postoperative; Hypersensitivity

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: The anesthetist is blinded to the arm of attribution
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Polyamine deficient diet (Experimental): Diet low in polyamines: the estimated calculated dose is 20 times lower that in an usual diet
  Interventions: Other: Polyamine Deficient Diet
- Control (No Intervention): Usual Diet plus two snacks

INTERVENTIONS:
Other: Polyamine Deficient Diet — Diet low in polyamines: the estimated calculated dose is 20 times lower that in an usual diet
  Arms: Polyamine deficient diet

SUMMARY:
The aim of this study is to evaluate if a polyamine deficient diet started 7 days prior to a major abdominal surgery (eventration cure and digestive continuity) and followed 7 days post-surgery reduces the area under the curve of the numerical pain rating scale in the 72 hours post-surgery.

DETAILED DESCRIPTION:
Morphine derivatives are known to be a major cause of postoperative ileus and also operative hyperalgesia. Operative hyperalgesia corresponds to an increase in morphine needs postoperatively which is proportional to the morphine dose necessary during the surgery. This effect is due to two mechanisms: opioids tolerance and induced hypersensitivity.

N-methyl-D-aspartate receptors (R-NMDA) play a key role in this induced hypersensitivity. Polyamines, organic compounds with several amines functions, are known R-NMDA agonists. They increase the phosphorylation of the tyrosine group within the NR2B subunit responsible for the inflammatory hyperalgesia.

Limiting the binding of polyamines to the R-NMDA seems an easy, safe and efficient way to limit the hypersensitivity induced post-operatively.

Most of the polyamines in the human body come from food. One study listed food regarding their polyamines content and allowed to check the safety of a polyamine deficient diet. Such a well-followed diet would allow to reduce by 20 the polyamines quantity present in the body.

The aim of this study is to evaluate whether a deficient polyamine diet introduced 7 days before and continued up to 7 days after an abdominal surgery requiring the use of morphine post-operatively reduces the post-operative pain, the consumption of analgesics (morphine) post-operatively and improve the recovery ability. Abdominals surgeries concerned will be the eventration cure and digestive continuity.

The medico-economic impact will be observed during this study.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years)
* Indication for a " major " abdominal surgery as second surgical procedure : cure of eventration and restoration of digestive continuity
* Intended Use of a Patient Controlled Morphine Pump (PCA) postoperatively or taking oral opioids
* Possible follow-up during 7 months (post-operative consultation at 1 month and 6 months only if postoperative pain or complications)
* Written informed consent form obtained from the patient
* Affiliated to the social security

Exclusion Criteria:

* Pregnant women
* Minor, adult under guardianship or benefiting from a legal protection
* Oncological surgery
* Surgery not painful (cholecystectomy, hernia, thyroidectomy, bariatric surgery)
* Drug addicts patients, or under opiate dependency
* Chronic pain patients (pain over 3 months)
* Patients in nursing home or convalescence home (diet non possible in institution)
* Planned hospitalisation before the intervention (during the 7 days before the surgery)
* Severe undernutrition defined by the HAS criteria (weight loss > 10% in 1 month and/or > 15% in 6 months, albumin at inclusion <15g/l)
* Patient refusing the possibility to change his eating habits
* Oral feeding impossible preoperatively
* Patient not able to express himself on their pain (silent, …)
* Decompensated psychiatric pathologies (severe depression syndrome,…)
* Patient unable to understand the protocol and/or to give his informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Estimated)
Dates: Start 2020-02-03 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
To show a 20% decrease of the area under the curve for the numerical pain rating scale in the 72 hours post-operative in the polyamine deficient diet group | 72 hours post-surgery
  To show a 20% decrease of the area under the curve for the numerical pain rating scale in the 72 hours post-operative in the polyamine deficient diet group measured every 6 hours in resting position, upon return from the operative room

SECONDARY OUTCOMES:
Change in the analgesics consumption post-operatively | 15 days post-surgery
  Measure of the analgesics consumption by the nurse during hospitalisation and by the patient with the patient book up to 15 days postsurgery
Change in the main dimension of pain | 6 months post-surgery
  Evaluation of the main dimension of pain using the Brief Pain Inventory (BPI)
Change of the recovery time of the gas transit | 6 months post-surgery
  Evaluation of the time to recover the gas transit post-surgery (in days)
Change of duration of urinary catheterization | 6 months post-surgery
  Recovery of spontaneous urination post-surgery (in days)
Change in the delay before the first postoperative lift | 6 months post-surgery
  Time before walking post-surgery (in days)
Change in length of hospitalisation stay and sick leave | 6 months post-surgery
  Hospitalisation time and sick leave (in days)
Change in neuropathic pain: Neuropathic pain scale (DN4) | 6 months post-surgery
  Use of the Neuropathic pain scale for patients seen for their postsurgery pain or complications. The scale contains 10 questions, the range is between 0-10, 10 being the worst score.
Change in global health status | 1 month before surgery, 1 month and 6 months post-surgery
  Use of autoquestionnaire EuroQol-5 Dimension (EQ-5D) to evaluate the global health status of the patients. The scale contains two parts, the first one contains 5 items to be completed by the patients with 5 levels for each item, the worst score being 55555. The second part is an analog visual scale with a range between 0-100, 0 being the worst score.
Change of the recovery ability | 1 month before surgery, 1 month and 6 months post-surgery
  Evaluation of the recovery ability using the Quality of Recovery-15 Questionnaire (QoR-15)
Change in the quality of life | 1 month before surgery, 1 month and 6 months post-surgery
  Assessment of the patient's quality of life by using the Short-Form Health Survey 36 questionnaire (SF-36)

CONTACTS AND LOCATIONS:
Overall Officials: Claire Blanchard, MD-PhD, Principal Investigator — Nantes University Hospital
Locations (4):
- France (4):
  - CHRU Brest La Cavale Blanche, Brest
  - Hôpital Louis Mourier from Ap-HP, Colombes
  - CHD Vendée, La Roche-sur-Yon
  - CHU Nantes Hôtel Dieu, Nantes